CLINICAL TRIAL: NCT06913556
Title: Comparing Effect of Hylorunic Acid and Lipid-coated Carbomer Gel on Dry Eyes After Phacoemulsification in Diabetic Patients
Brief Title: Comparing Effect of Hylorunic Acid and Lipid-coated Carbomer Gel on Dry Eyes After Phacoemulsification in DP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MSRSW/Batch-Fall23/807
Record Dates: First submitted 2025-03-29; First posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-03

CONDITIONS: Dry Eye Syndrome
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- preoperative dry eyes (Experimental)
  Interventions: Diagnostic Test: Preoperative dry eyes
- lipid coated carbomer gel eye drops (Experimental)
  Interventions: Combination Product: Lipid coated carbomer gel eye drops

INTERVENTIONS:
Diagnostic Test: Preoperative dry eyes — In group 1 we access preoperative dry eyes condition and postoperatively we access the condition in 2nd and 4th week with the use of Hylorunic acid lubricant.
  Arms: preoperative dry eyes
Combination Product: Lipid coated carbomer gel eye drops — In group 2 we prescribe the lipid coated carbomer gel eye drops and access dry eyes condition preoperative and postoperative on 2nd and 4th week and check the curative effect of drop.
  Arms: lipid coated carbomer gel eye drops

SUMMARY:
In this research checked the curative effect of two different artificial tears on dry eyes after phacoemulsification was checked. In research, the randomized control trial methodology is used

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 50-70
* Both gender male /female

Exclusion Criteria:

* Patients who have acute dry eye condition before phacoemulsification cataract surgery.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2025-03-20 (Actual); Primary Completion 2025-06-20 (Estimated); Study Completion 2026-02-20 (Estimated)

PRIMARY OUTCOMES:
The Tear Break-Up Time (TBUT) test | 12 Months
  The Tear Break-Up Time (TBUT) test measures how long the tear film on the eye surface remains intact before it breaks up, with a normal TBUT typically being 10 seconds or more. A shorter TBUT suggests tear film instability and potential dry eye issues.
Schirmer test | 12 Months
  In a Schirmer test, a score of greater than 10 mm of moistened area on the filter paper after 5 minutes is considered normal, while less than 10 mm suggests dry eyes

CONTACTS AND LOCATIONS:
Locations (1):
- Shaheen welfare hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No